CLINICAL TRIAL: NCT01333839
Title: Impact of CABG Surgery and Subsequent Exercise Intervention on Insulin Sensitivity and Muscle Mass: a Cluster Randomized Trial
Brief Title: Impact of Coronary Artery Bypass Graft (CABG) Surgery on Skeletal Muscle Mass and Insulin Sensitivity, Followed by Exercise Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, Dominique Hansen, Associate Professor, Hasselt University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CABG2011
Record Dates: First submitted 2011-04-06; First posted 2011-04-12 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Coronary Artery Disease
Keywords: CABG surgery; exercise intervention; insulin sensitivity; muscle mass
MeSH Terms: conditions — Coronary Artery Disease; Insulin Resistance | interventions — Exercise; Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- standard exercise intervention (Active Comparator): 12 weeks of endurance exercise training
  Interventions: Other: exercise training
- modified exercise intervention (Active Comparator): combined endurance + strength exercise training
  Interventions: Other: exercise training
- modified 2 exercise intervention (Active Comparator): combined endurance + strength exercise training + oral protein supplements
  Interventions: Other: exercise training

INTERVENTIONS:
Other: exercise training — endurance exercise training: 40 min of exercise at 65% of VO2peak, 3 days/week
  Other Names: Rehabilitation

SUMMARY:
In this study, the investigators want to examine the impact of coronary artery bypass graft (CABG) surgery on skeletal muscle mass, muscle metabolism, and insulin sensitivity in 90 subjects. In extent, the impact of a subsequent exercise intervention will be examined, with a follow-up up to 12 months after surgery.

DETAILED DESCRIPTION:
90 subjects undergoing elective CABG surgery will be included. These subjects are free from orthopedic limitations, will have no severe complications during surgery, and are willing to participate in a 12-week exercise training intervention.

At baseline (before surgery), following parameters will be assessed: blood parameters (glycemic control, lipid profile, anabolic/catabolic hormones, inflammatory markers), body composition (by dual x-ray absorptiometry), handgrip strength, and general subject features (medication, gender, age, etc.).

The first three days after surgery, blood samples will be collected for the analysis of glycemic control, lipid profile, anabolic/catabolic hormones, inflammatory markers.

Next, at the start of exercise intervention, after 6 and 12 weeks of exercise training, and after a 12-month follow-up, following parameters will be assessed: blood parameters (glycemic control, lipid profile, anabolic/catabolic hormones, inflammatory markers), body composition (by dual x-ray absorptiometry), handgrip strength, maximal exercise capacity (by ergospirometry testing), physical activity (by questionnaire), and quality of life ( by questionnaire).

At 12 months of follow-up, cardiovascular mortality and morbidity (re-occurrence of angina, acute myocardial infarction, need for surgery, death) will be assessed.

When initiating exercise intervention, subjects will randomly (n=30 in each group) be assigned to 12 weeks of standard exercise intervention (endurance exercise training), modified exercise intervention (endurance exercise training + strength training), or modified exercise intervention (endurance exercise training + strength training + oral protein supplements).

This will be a cluster randomized clinical trial. Investigators executing the measurements will be blinded for treatment allocation.

ELIGIBILITY:
Inclusion Criteria:

* Elective CABG surgery
* Willing to participate in 12-week exercise intervention

Exclusion Criteria:

* Complicated surgery
* Severe complications during first days after CABG surgery
* Orthopedic limitations that interfere with proper exercise intervention participation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-02; Primary Completion 2015-02 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
change in muscle mass and insulin sensitivity | pre-operative, 1, 2, 3 days, and 2, 12, 54 weeks after surgery
  Baseline insulin sensitivity and muscle mass will be assessed ahead of surgery. Afterwards, the change in these parameters will be assessed at various predefined timepoints.

SECONDARY OUTCOMES:
change in exercise capacity | 2, 12, 54 weeks after surgery
  Baseline exercise capacity will be assessed at 2 weeks after surgery. Afterwards, the change in this parameters will be assessed at various predefined timepoints.

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Hansen, PhD, Principal Investigator — Jessa Hospital, Hasselt, Belgium
Locations (1):
- Jessa Hospital, Hasselt, Belgium